CLINICAL TRIAL: NCT01562080
Title: Combined Effects of Bioactive Compounds (ARMOLIPID PLUS ®) on Lipid Profile and Clinical Criteria of Metabolic Syndrome in Patients With Serum Elevated LDL-C
Brief Title: Combined Effects of Bioactive Compounds in Lipid Profile
Acronym: ARM-PLUS-LDL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Collaborators: Centro Tecnológico de Nutrición y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARM-PLUS-LDL
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Hyperlipidemia; Low-density-lipoprotein-type; Elevated Triglycerides
Keywords: hyperlipidemia; metabolic syndrome; yeast red; berberine; policosanol; astaxanthin
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement (Experimental): red yeast, astaxanthin, berberine, policosanol, coenzyme Q10, folic acid
  Interventions: Dietary Supplement: Armolipid Plus
- microcrystalline cellulose (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Armolipid Plus — one tablet per day during 12 weeks
  Arms: Dietary supplement
Dietary Supplement: placebo — one tablet per day during 12 weeks
  Arms: microcrystalline cellulose

SUMMARY:
The aim of this study is to demonstrate whether, along with dietary recommendations, Armolipid Plus ® can improve the profile of patients with elevated plasma LDL-C acting as a change of lifestyle therapy (TLC) according to the definition of Adult Treatment Panel III (ATP III)

DETAILED DESCRIPTION:
Recently reported that the combination of extract of red yeast rice policosanol composed, berberine, folic acid and coenzyme Q10 (Armolipid Plus ®, Rottapharm) produced a significant improvement in lipid profile in patients with moderately elevated cholesterol levels of low density lipoprotein (LDL-C) plasma.

Taking into account the potential effect of Armolipid Plus ® on the lipid profile, it is important to investigate the effectiveness in the field of cardiovascular prevention to define its position in prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years old
* LDL-c plasma levels ≥130 mg/dL and ≤ 189 mg/dL
* Patients not requiring lipid-lowering drug treatment according to ATPIII guidelines,that do not have cardiovascular disease, stroke or intermittent claudication, diabetes mellitus, renal or Patients who have demonstrated effects or contraindications to lipid-lowering drug therapy (in this case, treatment should be discontinued 1 month before baseline.
* Signed and dated informed consent before any study specific procedure.

Exclusion Criteria:

* Patients on drug therapy to reduce LDL-C, for example, statins, bile acid sequestrants, nicotinic acid, fibrates or similar (up to 1 month before baseline).
* History of cardiovascular disease, stroke or intermittent claudication.
* Diabetes mellitus (at least 2 blood fasting glucose greater than 126 mg / dL).
* Having taken any functional food with sterols, stanols or similar or any nutraceutical with lipid-lowering effects during the previous 7 days.
* Plasma levels of triglycerides > 350 mg/dl
* Diagnosis of familial hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
investigate whether the addition of Armolipid Plus ® decreases by 20% LDL-C levels compared to baseline in patients with initial levels of LDL-C ≥ 130 mg / dL. | twelve weeks

SECONDARY OUTCOMES:
Cardiovascular risk (according to the Framingham tables). | twelve weeks
Criteria for Metabolic Syndrome | twelve weeks
Levels of triglycerides and cholesterol high density lipoprotein (HDL-C). | twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, MD PhD, Study Director — Hosp. Universitari Sant Joan de Reus (Tarragona); Jesús Millán, MD PhD, Principal Investigator — Hosp. Universitario Gregorio Marañón (Madrid); José R Calabuig, MD PhD, Principal Investigator — Hosp. Universitario La Fe (Valencia); José Villar, MD PhD, Principal Investigator — Hosp. Universitario Virgen del Rocío (Sevilla); José Puzo, MD PhD, Principal Investigator — Hosp. Universitario San Jorge (Huesca); Angel Brea, MD, Principal Investigator — Hosp. Universitario San Pedro ( Logroño)
Locations (1):
- Hosp. Universitario San Joan, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Sola R, Valls RM, Puzo J, Calabuig JR, Brea A, Pedret A, Morina D, Villar J, Millan J, Anguera A. Effects of poly-bioactive compounds on lipid profile and body weight in a moderately hypercholesterolemic population with low cardiovascular disease risk: a multicenter randomized trial. PLoS One. 2014 Aug 1;9(8):e101978. doi: 10.1371/journal.pone.0101978. eCollection 2014. PMID 25084280